CLINICAL TRIAL: NCT04032327
Title: Efficacy of Injectable Local Anesthetics on Postsurgical Analgesia Following Posterior Colporrhaphy: A Prospective, Randomized, Double-Blinded Trial
Brief Title: Local Anesthetics on Postsurgical Analgesia Following Posterior Colporrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Dengler, MD, FPMRS Fellow, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2018-03-27; First posted 2019-07-25 (Actual); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Plain Bupivacaine (Active Comparator): 20 mL of 0.25% plain bupivacaine
  Interventions: Drug: Bupivacaine
- Exparel plus plain bupivacaine (Active Comparator): 10 mL of extended release liposomal bupivacaine (Exparel) plus 10 mL of 0.25% plain bupivacaine mixed
  Interventions: Drug: Exparel plus plain bupivacaine

INTERVENTIONS:
Drug: Exparel plus plain bupivacaine — 10 mL of extended release liposomal bupivacaine (Exparel) plus 10 mL of 0.25% plain bupivacaine mixed to be injected vaginally prior to the start of posterior colporrhaphy
  Other Names: extended release liposomal bupivacaine plus marcaine
  Arms: Exparel plus plain bupivacaine
Drug: Bupivacaine — 20 mL of 0.25% plain bupivacaine to be injected vaginally prior to the start of posterior colporrhaphy
  Other Names: marcaine
  Arms: Plain Bupivacaine

SUMMARY:
Effective post-surgical pain management is a crucial component of a patient's postoperative course following posterior colporrhaphy. Narcotics are the cornerstone for postoperative analgesia with a frequent re-dosing requirement, a lengthy list of side effects and adverse reaction risks. The colorectal, orthopedic and general surgery literatures have reported on an extended-release bupivacaine liposomal injection, Exparel®, which remarkably reduces acute post-operative pain; however, literature regarding this medication specific to Urogynecology and Gynecology is limited.

The investigators propose a prospective, randomized, double blind, trial with 120 subjects recruited from the Walter Reed National Military Medical Center (WRNMMC) Urogynecology Clinic to study postsurgical pain control after posterior repair. There will be two arms in the study; one arm with bupivacaine alone and a second arm with bupivacaine mixed with Exparel®(extended-release, liposomal bupivacaine) injected vaginally in patients undergoing posterior colporrhaphy. Subjects will be randomized to receive either 20 milliliter (mL) of plain bupivacaine or 20mL (10ml+10ml) mixture of bupivacaine plus Exparel®.

The primary objective of the trial will be to evaluate the postsurgical vaginal pain using a visual analog pain scale at days 1, 2, 3 post-procedure. All subjects will have acetaminophen, a non-steroidal anti-inflammatory drug and narcotic pain medication available for pain control regardless of assignment, which is the usual postoperative pain control regimen. The investigators hypothesize a 30% difference in post-operative pain measurements between the two groups.

Additional objectives of this study are to evaluate total medication usage on days 1, 2 and 3 and any post-operative voiding and defecatory dysfunction, comparing the two groups

ELIGIBILITY:
Inclusion Criteria:

* Females >18 years of age undergoing Urogynecologic surgery involving the posterior vaginal wall mucosa or muscularis including posterior colporrhaphy at Walter Reed National Military Medical Center.
* Patients must be able to read and understand written English or have an appropriate certified medical translator available.

Exclusion Criteria:

* Known allergy to amide local anesthetics.
* Unstable cardiac arrhythmia.
* Hepatic impairment (including but not limited to patients under the care of their physician for severe hepatic disease, cirrhosis or hepatic cancer).
* Known pregnancy at time of surgery (pregnancy test morning of surgery if applicable).
* Regular use of narcotic pain medication, defined as use on most days of week at any time in the three months prior to surgery.
* Significant history of opioid or alcohol abuse or addiction (requiring treatment).
* Concurrent pain management requiring the use of epidural anesthesia.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females only
Enrollment: 120 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gruber, MD, Study Chair — Walter Reed National Military Medical Center (WRNMMC)
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dengler KL, Craig ER, DiCarlo-Meacham AM, Welch EK, Brooks DI, Vaccaro CM, Gruber DD. Preoperative pudendal block with liposomal and plain bupivacaine reduces pain associated with posterior colporrhaphy: a double-blinded, randomized controlled trial. Am J Obstet Gynecol. 2021 Nov;225(5):556.e1-556.e10. doi: 10.1016/j.ajog.2021.08.034. Epub 2021 Aug 30. PMID 34473963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The two populations were analyzed separately.
  years
    Plain Bupivacaine: number analyzed (Participants) | 60 | 0 | 60
    Plain Bupivacaine | 49.5 [40.0 to 61.0] |  | 49.5 [40.0 to 61.0]
    Exparel Plus Plain Bupivacaine: number analyzed (Participants) | 0 | 60 | 60
    Exparel Plus Plain Bupivacaine |  | 51.0 [42.8 to 62.0] | 51.0 [42.8 to 62.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 46 | 48 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: The two populations were analyzed separately.
  kg/m^2
    Plain Bupivacaine: number analyzed (Participants) | 60 | 0 | 60
    Plain Bupivacaine | 26.1 [23.7 to 30.3] |  | 26.1 [23.7 to 30.3]
    Exparel plus plain bupivacaine: number analyzed (Participants) | 0 | 60 | 60
    Exparel plus plain bupivacaine |  | 25.9 [23.3 to 31.0] | 25.9 [23.3 to 31.0]
Gravidity [Median (Inter-Quartile Range); unit: pregnancies] — Population: The two populations were analyzed separately.
  pregnancies
    Plain Bupivacaine: number analyzed (Participants) | 60 | 0 | 60
    Plain Bupivacaine | 3 [2 to 3] |  | 3 [2 to 3]
    Exparel plus plain bupivacaine: number analyzed (Participants) | 0 | 60 | 60
    Exparel plus plain bupivacaine |  | 3 [2 to 4] | 3 [2 to 4]
Parity [Median (Inter-Quartile Range); unit: births] — Population: The two populations were analyzed separately.
  births
    Plain Bupivacaine: number analyzed (Participants) | 60 | 0 | 60
    Plain Bupivacaine | 2 [2 to 3] |  | 2 [2 to 3]
    Exparel plus plain bupivacaine: number analyzed (Participants) | 0 | 60 | 60
    Exparel plus plain bupivacaine |  | 3 [2 to 3] | 3 [2 to 3]
colpopexy [Count of Participants; unit: Participants]
  none | 12 | 9 | 21
  laparoscopic | 32 | 31 | 63
  vaginal | 16 | 20 | 36
hysterectomy [Count of Participants; unit: Participants]
  none | 21 | 25 | 46
  laparoscopic | 30 | 22 | 52
  vaginal | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Vaginal Pain Scores Using the Defense and Veterans Pain Rating Scale (Visual Analog Scale) Between Bupivacaine Alone Versus Exparel® Following Posterior Colporrhaphy Post-operatively
Description: Patients will be asked on postoperative day (POD) 1 to provide numerical values regarding vaginal pain from 0-10 (zero being no pain and 10 being the worst pain) utilizing the Defense and Veterans Pain Rating Scale (visual analog scale)
Time Frame: Subjects will be asked to provide numerical values on postoperative day 1.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 2 [0 to 4] | 0 [0 to 2]

2. Primary Outcome: Change in Vaginal Pain Scores Using the Defense and Veterans Pain Rating Scale (Visual Analog Scale) Between Bupivacaine Alone Versus Exparel® Following Posterior Colporrhaphy Post-operatively
Description: Patients will be asked on postoperative day (POD) 2 to provide numerical values for vaginal pain from 0-10 (zero being no pain and 10 being the worst pain) utilizing the Defense and Veterans Pain Rating Scale (visual analog scale)
Time Frame: Subjects will be asked to provide numerical values on postoperative day 2.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 3 [2 to 5] | 2 [1 to 4]

3. Primary Outcome: Change in Vaginal Pain Scores Using the Defense and Veterans Pain Rating Scale (Visual Analog Scale) Between Bupivacaine Alone Versus Exparel® Following Posterior Colporrhaphy Post-operatively
Description: Patients will be asked on postoperative day (POD) 3 to provide numerical values for vaginal pain from 0-10 (zero being no pain and 10 being the worst pain) utilizing the Defense and Veterans Pain Rating Scale (visual analog scale)
Time Frame: Subjects will be asked to provide numerical values on postoperative day 3.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 3 [2 to 5] | 2 [1 to 4]

4. Secondary Outcome: Amount Ibuprofen Pain Medication Required During the Postoperative Period at Home
Description: Calculate total postoperative ibuprofen used while at home via perform pill counts on postoperative days 1, 2, 3 (done via a phone call). This will allow calculation of total amount of ibuprofen utilized at home through postoperative day #3
Time Frame: Calculated with phone call on postoperative day 1, 2, and 3 (total acetaminophen utilized at home)
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
milligrams | 3600 [2400 to 4800] | 2400 [0 to 4050]

5. Secondary Outcome: Amount Acetaminophen Pain Medication Required During the Postoperative Period at Home
Description: Calculate total postoperative acetaminophen used while at home via perform pill counts on postoperative days 1, 2, 3 (done via a phone call). This will allow calculation of total amount of acetaminophen utilized at home through postoperative day #3
Time Frame: Calculated with phone call on postoperative day 1, 2, and 3 (total acetaminophen utilized at home)
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
milligrams | 4000 [2110 to 5930] | 3250 [1300 to 4550]

6. Secondary Outcome: Amount Opioid Pain Medication Required During the Postoperative Period (Through Day 3)
Description: Calculate total postoperative opioid medications used while inpatient and perform pill counts on postoperative days 1, 2, 3 (done via a phone call or inpatient). This will allow calculation of total amount of opioid pain medications utilized through postoperative day #3
Time Frame: Calculated throughout hospitalization and/or with phone call on postoperative day 1, 2, and 3 (total opioids utilized)
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
morphine milligram equivalents | 45.0 [22.5 to 118] | 57.1 [30.0 to 93.5]

7. Secondary Outcome: Percentage of Participants Who Passed Active Voiding Trial Comparing the Bupivacaine Plus Exparel® Group Versus the Bupivacaine Plain Group.
Description: Investigators will record in patients passed active voiding trail prior to discharge home.
Time Frame: Postoperative active voiding trial on postoperative day 1.
Measure: Number; unit: percentage passed
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
percentage passed | 82 | 72

8. Secondary Outcome: Rate of Post-operative Defecatory Function After Posterior Colporrhaphy, Comparing the Bupivacaine Plus Exparel® Group Versus the Bupivacaine Plain Group.
Description: Investigators will record in patients have had a bowel movement within the first three days postoperatively.
Time Frame: Postoperatively up to day 3
Measure: Number; unit: percentage of patients
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
percentage of patients | 71.6 | 73.3

9. Secondary Outcome: Impact of Vaginal Pain Scores on Quality of Life Measures (ACTIVITY) Using Defense and Veterans Pain Rating Scale (Visual Analog Scale) Comparing the Bupivacaine Plus Exparel® Group and the Bupivacaine Plain Group
Description: Investigators will ask patients "how is your vaginal pain impacting your ACTIVITY (quality of life question)" and respond using a 0-10 answer (0 being no impact and 10 being significant impact) using the Defense and Veterans Pain Rating Scale (visual analog scale). This will be recorded on POD 3
Time Frame: Subjects will be asked to provide numerical value on postoperative day 3.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 3.5 [0.250 to 6] | 3 [0.500 to 5]

10. Secondary Outcome: Impact of Vaginal Pain Scores on Quality of Life Measure (SLEEP) Using Defense and Veterans Pain Rating Scale (Visual Analog Scale) Comparing the Bupivacaine Plus Exparel® Group and the Bupivacaine Plain Group
Description: Investigators will ask patients "how is your vaginal pain impacting your SLEEP (quality of life question)" and respond using a 0-10 answer (0 being no impact and 10 being significant impact) using the Defense and Veterans Pain Rating Scale (visual analog scale). This will be recorded on POD 3
Time Frame: Subjects will be asked to provide numerical value on postoperative day 3.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 0.500 [0 to 3] | 1 [0 to 3]

11. Secondary Outcome: Impact of Vaginal Pain Scores on Quality of Life Measure (MOOD) Using Defense and Veterans Pain Rating Scale (Visual Analog Scale) Comparing the Bupivacaine Plus Exparel® Group and the Bupivacaine Plain Group
Description: Investigators will ask patients "how is your vaginal pain impacting your MOOD (quality of life question)" and respond using a 0-10 answer (0 being no impact and 10 being significant impact) using the Defense and Veterans Pain Rating Scale (visual analog scale). This will be recorded on POD 3
Time Frame: Subjects will be asked to provide numerical value on postoperative day 3.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 1 [0 to 3] | 1 [0 to 3]

12. Secondary Outcome: Impact of Vaginal Pain Scores on Quality of Life Measure (STRESS) Using Defense and Veterans Pain Rating Scale (Visual Analog Scale) Comparing the Bupivacaine Plus Exparel® Group and the Bupivacaine Plain Group
Description: Investigators will ask patients "how is your vaginal pain impacting your STRESS (quality of life question)" and respond using a 0-10 answer (0 being no impact and 10 being significant impact) using the Defense and Veterans Pain Rating Scale (visual analog scale). This will be recorded on POD 3
Time Frame: Subjects will be asked to provide numerical value on postoperative day 3.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
Number analyzed (Participants) | 60 | 60
score on a scale | 0 [0 to 3] | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: entirety of the study (AUG2018-AUG2020); patients were followed out to 6 weeks postoperatively
Arm/Group | Plain Bupivacaine | Exparel Plus Plain Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 3/60 | 4/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plain Bupivacaine (N=60) | Exparel Plus Plain Bupivacaine (N=60)
Postoperative sensory numbness/tingling in the lower extremities (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04032327/Prot_SAP_ICF_001.pdf